CLINICAL TRIAL: NCT06921538
Title: A Novel Home-based Non-invasive Neuromodulation Therapy for Children and Adolescents With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Ng Zhi Min, Principal Investigator, KK Women's and Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024/00201
Record Dates: First submitted 2024-11-18; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy (CP)
Keywords: neuromodulation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Intervention is non-invasive neuromodulation device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: Standard care + AscenZ-IV Stimulation (Experimental): Participants randomized as Group 1 first receive both standard care (existing medical interventions, therapy program) and AscenZ-IV Stimulation for 8 weeks (30min/day; 5 to 7 sessions/week, additional 30min/day; 5 to 7 sessions/week for behavioral and drooling issues if necessary). Then, they receive standard care only for another 8 weeks. For participants randomized as Group 2, control condition precedes intervention condition. Subsequently, participants are given the option to receive an additional 4 weeks of intervention for maintenance
  Interventions: Device: AscenZ-IV neuromodulation device
- Control: Standard care only (No Intervention): Participants randomized as Group 1 first receive both standard care (existing medical interventions, therapy program) and AscenZ-IV Stimulation for 8 weeks (30min/day; 5 to 7 sessions/week, additional 30min/day; 5 to 7 sessions/week for behavioral and drooling issues if necessary). Then, they receive standard care only for another 8 weeks. For participants randomized as Group 2, control condition precedes intervention condition. Subsequently, participants are given the option to receive an additional 4 weeks of intervention for maintenance

INTERVENTIONS:
Device: AscenZ-IV neuromodulation device — AscenZ-IV neuromodulation device is a novel treatment modality that utilizes 2 non-invasive neuromodulation technologies - tPCS and TENS - concurrently within a device. The home-based, non-invasive AscenZ-IV Stimulator therapy has been shown to improve spasticity and motor function
  Arms: Intervention: Standard care + AscenZ-IV Stimulation

SUMMARY:
The aim of this study is to evaluate the clinical effectiveness, feasibility and acceptability of a novel home-based noninvasive neuromodulation therapy (AscenZ-IV Stimulator) that utilizes transcranial Pulse Current Stimulation (tPCS) and Transcutaneous Electrical Nerve Stimulation (TENS) for children and adolescents with cerebral palsy as a community-based intervention by families and healthcare providers.

DETAILED DESCRIPTION:
Currently there is no cure for CP, with treatments limited to oral medications, physical therapies, splinting and casting, botulinum toxin injections and invasive surgical methods. These approaches are time-consuming, labor-intensive and are associated with high direct and indirect costs which reduce patient adherence over the long term. Some are invasive, short-lasting and associated with high risks. Likewise, there is an unmet clinical need for an alternative therapy that can effectively reduce spasticity and improve motor function while being non-invasive, less labor-intensive, affordable and homebased, with minimal side-effects.

The AscenZ-IV neuromodulation device is a novel treatment modality that utilizes 2 non-invasive neuromodulation technologies - tPCS and TENS - concurrently within a device. The home-based, non-invasive AscenZ-IV Stimulator therapy has been shown to improve spasticity and motor function, as well as reduce direct and indirect costs in China (unpublished). The stimulator is HSA-approved for children aged 2 to 12. This study includes children and adolescents with mild to severe Spastic Cerebral Palsy (CP) from age 2 to <21 and Gross Motor Function Classification System (GMFCS) II, III, IV, V.

The hypothesis of this crossover randomized controlled trial is that the application of the AscenZ-IV neuromodulation device is an effective and cost-effective home-based, caregiver-delivered adjunct therapy for children with CP to improve their spasticity, motor function and quality of life.

The study is designed as a mixed method approach consisting of a crossover randomized controlled trial, as well as questionnaires and medical records. The former is to compare between standard care (existing medical interventions, therapy program) and intervention (standard care + AscenZ-IV stimulation for 8 weeks) by performing physical and functional assessments. The latter is to understand the key barriers and facilitators for adoption of the AscenZ-IV stimulator for CP.

ELIGIBILITY:
Inclusion Criteria:

Children and adolescents aged between 2 to <21 years old with mild to severe Spastic Cerebral Palsy (CP) classified on Gross Motor Function Classification System (GMFCS) II, III, IV, V. Families with at least one parent or caregiver has simple or conversational English language skill.

To be eligible for the qualitative interview components of this research study, the individuals should be recognised as one of the following:

1. CP patients who participate in this research study,
2. caregivers of the CP patients taking part in this research study,
3. implementation staff
4. qualified clinicians not involved in the intervention or refused to recommend the intervention device (AscenZion-IV stimulator) for management of CP.

Eligible individuals must agree to be audio-recorded.

Exclusion Criteria:

1. CP patients with epilepsy with recent seizures (<12 months) will be excluded for safety given the theoretical risks of seizures (abnormal brain electrical discharges) with transcranial electrical stimulation. We will include those with well controlled epilepsy with no recent seizures (within 12 months).
2. CP patients who have contra-indications to the use of tPCS and/or TENS will be excluded from the study, include:

   * Individuals with history of uncontrolled epileptic disorder, seizures, brain tumour or trauma, and mental disease
   * Individuals with electrical implanted stimulatory device, such as pacemaker or defibrillator
   * Individuals with medical devices that are affected by magnets, such as programmable shunts.
   * Individuals with pregnancy
3. CP patients who received any intramuscular botulinum toxin injections within less than 6 months (as anti-spasticity effect lasts for 4-6 months).
4. CP patients who received any musculo-skeletal, brain or nerve-related surgery within less than 6 months, or major surgery requiring prolonged hospitalisation (>1week) within less than 3 months.

Those who do not agree to be audio-recorded will be excluded for the qualitative interview components of this research study.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Spasticity | At baseline, at Week 8 and Week 16 of the crossover design, and final assessments i.e. Week 20 after the maintenance phase.
  Physical assessments using the Modified Tardieu Scale (MTS) for upper and/or lower limbs are performed to assess improvement in spasticity with the aim of reducing the R2-R1 value. R1 refers to 'first catch or resistance' or the angle at which there is initial resistance when the muscle is stretched passively. R2 refers to 'end range resistance' or the angle at which the muscle reaches full range of motion under passive stretch, where resistance decreases or disappears. Min (R2-R1) = 0° indicates no spasticity (better outcome); Max (R2-R1) = 90° indicates severe spasticity (worse outcome).

SECONDARY OUTCOMES:
Gross Motor Function | At baseline, at Week 8 and Week 16 of the crossover design, and final assessments i.e. Week 20 after the maintenance phase.
  Improvement in gross motor function for CP patients is assessed using the Gross Motor Function Measure 66 (GMFM-66) score. Scoring is based on a 4-point scale (0 - does not initiate, 1 - initiates, 2 - partially completes, 3 - completes, NT - not tested) for each of the 66 items. The minimum GMFM-66 score is 0 (worse outcome), which indicates that the child is unable to perform any of the tasks in the assessment. The maximum GMFM-66 score is 100 (better outcome), which indicates that the child can perform all tasks to the full extent expected for their age.
Upper Limb Motor Function | At baseline, at Week 8 and Week 16 of the crossover design, and final assessments i.e. Week 20 after the maintenance phase.
  Improvement in manual ability for children with upper limb impairments is assessed using the ABILHAND-Kids assessment composed of 21 assessment items, each scored on a 3-point scale (Impossible, Difficult, Easy). The raw score is undergone Rasch conversion to get a global score ranging from 0 to 40. A higher score indicates better manual ability. ABILHAND-Kids is only assessed for participants with hemi/quadriplegia and MACS I to III.
Gait Function | At baseline, at Week 8 and Week 16 of the crossover design, and final assessments i.e. Week 20 after the maintenance phase.
  The Gait Outcomes Assessment List (GOAL) is used to assess the quality of walking and how it impacts daily life and mobility. Assessment items include activities of daily living and independence, gait function and mobility, pain, discomfort and fatigue, physical activities, sport and recreation, gait pattern and appearance, as well as use of braces and mobility aids. Each item is scored from 0 (severe limitation) to 5 (no limitation), or 0 (very unhappy) to 4 (very happy), thus giving a total score ranging from 0 (severe limitations in all areas) to maximum 236 (no limitation or optimal walking function in all areas). GOAL is only assessed for CP patients of GMFCS II or III.
Cerebral Palsy-specific Health-related Quality of Life | At baseline, at Week 8 and Week 16 of the crossover design, and final assessments i.e. Week 20 after the maintenance phase.
  Cerebral Palsy-specific Health-related Quality of Life is assessed using the Pediatric Quality of Life Inventory™ 3.0 Cerebral Palsy Module (PedsQL™ 3.0 Cerebral Palsy Module). Items are measured on a 5-point Likert scale from 0 (Never a problem) to 4 (Almost always a problem). Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Scores are transformed to a 1 to 100 scale. Higher scores indicate lower problems thus better cerebral palsy-specific health-related quality of life.
General Health-related Quality of Life | At baseline, at Week 8 and Week 16 of the crossover design, and final assessments i.e. Week 20 after the maintenance phase.
  General health-related quality of life is assessed using EQ-5D-Y-3L. The items assess 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. There are 3 possible response levels for each dimension - level 1 (no problem), level 2 (some problems), level 3 (a lot of problems). The minimum total score is represented as 11111 on the index, indicating best health state. The maximum total score is represented as 33333 on the index, indicating worst health state.
Quality of Life - Care and Comfort | At baseline, at Week 8 and Week 16 of the crossover design, and final assessments i.e. Week 20 after the maintenance phase.
  The ICF-8 items for Care and Comfort is part of the International Classification of Functioning, Disability and Health (ICF) framework. 8 items have been selected, 2 of which assess quality of life in terms of activities and participation, scored from 0 = no difficulty to 4 = complete difficulty. The other 6 items assess quality of life in terms of body function, scored from 0 = no impairment to 4 = complete impairment. The total minimum score is 0 indicating no difficulty and impairment, thus high quality of life, whereas the maximum score is 32 indicating complete difficulty and impairment, thus poor quality of life. ICF-8 is assessed only for subjects with dystonia.

OTHER OUTCOMES:
Drooling | At baseline, at Week 8 and Week 16 of the crossover design, and final assessments i.e. Week 20 after the maintenance phase
  Daniel Drooling Impact Scale Questionnaire (DDISQ) is used to assess reduction of drooling. The 20-item questionnaire was designed with responses scored on a 5-point scale with increasing quantity or severity in impact (in a consistent manner). The summated score will be used for analysis and interpretation. A higher value represents a worse outcome.
Behavior | At baseline, at Week 8 and Week 16 of the crossover design, and final assessments i.e. Week 20 after the maintenance phase
  For participants with behavioral issues, the Aberrant Behavior Checklist is to assess improvement in behavior. The ABC comprises 58 items scored on a 4-point Likert scale (0 = no problem, 1 = minor problem, 2 = moderate problem, 3 = severe problem). Item scores are additive, and higher scores reflect more severe levels of challenging behaviour.
Dystonia Severity | At baseline, at Week 8 and Week 16 of the crossover design, and final assessments i.e. Week 20 after the maintenance phase
  For participants with dystonia, the Dystonia Severity Action Plan (DSAP) is used to assess reduction of dystonia. Grade 1 to 5 - Severity increases as the grade increases.
Estimated Patient Cost | At baseline, at Week 8 and Week 16 of the crossover design, and final assessments i.e. Week 20 after the maintenance phase
  Cost effectiveness of the device is assessed using the economic evaluation forms at baseline and post-intervention, as well as medical records. Data collected include direct medical costs outside of the hospital (ex. private health services) as well as direct non-medical costs (ex. home modifications, equipment, etc.), indirect costs (ex. lost productivity) and willingness to pay. A higher cost indicates larger burden to the patient, thus worse outcome.
Patient and Caregivers' Satisfaction | At baseline, at Week 8 and Week 16 of the crossover design, and final assessments i.e. Week 20 after the maintenance phase
  Patient and caregivers' device satisfaction measures are assessed using the Usability-5D questionnaire. From a score scale from 1 (totally disagree) to 7 (totally agree) the effectiveness, error tolerance, practicality, level of engagement, etc. and overall experience of using the device will be assessed. Lower score indicates lower satisfaction and higher score indicates higher satisfaction. Qualitative data is also captured, for whether they are keen to try the device again (yes/no). The questionnaire items will be analyzed and reported descriptively.
Stakeholder Acceptability | At baseline, at Week 8 and Week 16 of the crossover design, and final assessments i.e. Week 20 after the maintenance phase
  Acceptability by stakeholders is assessed using the Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM) questionnaire. The questionnaire consists of 4 items in each category measured on a 5-point Likert scale from 1 (Completely disagree) to 5 (Completely agree). Scales can be created for each measure by averaging responses. Scale values range from 1 to 5. Higher scores indicate greater acceptability, appropriateness, or feasibility, thus better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Min Ng, MBBS, MRCPCH, Principal Investigator — KK Women's and Children's Hospital; Jeremy Lin, MBBS, MRCPCH, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital Singapore, Singapore
  - KK Women's and Children's Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No
Not approved to share IPD